CLINICAL TRIAL: NCT06156579
Title: Phase II Study of (Early) Combination Salvage Therapy With Venetoclax and Intensified Decitabine in Relapsed/Refractory AML
Brief Title: Combination Salvage Therapy With Venetoclax and Decitabine in Relapsed/Refractory AML
Acronym: VenSwitch
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VenSwitch
Record Dates: First submitted 2023-11-13; First posted 2023-12-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-12

CONDITIONS: AML; MDS
Keywords: Venetoclax; Decitabine; salvage therapy
MeSH Terms: interventions — Decitabine; venetoclax

STUDY DESIGN:
Intervention Model Description: single center, one arm, open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Salvage therapy with Venetoclax and intensified Decitabine
  Interventions: Drug: Decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine — Decitabine 20 mg/m^2, i.v., once daily, 10 days
  Other Names: Dacogen
Drug: Venetoclax — Venetoclax, 400 mg, p.o., once daily, 28 days
  Other Names: Venclyxto; Venclexta

SUMMARY:
The goal of this prospective, phase II single center, one arm, open label clinical trial is to test the efficacy and feasibility of a combination salvage therapy with Venetoclax and intensified Decitabine in patients with newly diagnosed AML (acute myeloid leukemia) and primary induction failure and patients with relapse of AML/MDS IB2 (myelodysplastic neoplasm with increased blasts 2) after chemotherapy. The primary endpoint is hematologic remission after treatment with Decitabine and Venetoclax. Participants eligible for the trial will receive a treatment of ten days of Decitabine and twenty-eight days of Venetoclax for one or two cycles, after which hematological remission will be assessed. Follow up will include the first one hundred days after end of treatment.

DETAILED DESCRIPTION:
This is a prospective, phase II single center one arm, open label clinical trial testing the efficacy and feasibility of a combination salvage therapy with Venetoclax and intensified Decitabine in relapsed or refractory AML and MDS IB2. Enrolled will be twenty-seven patients with newly diagnosed AML and primary induction failure to conventional anthracycline-based induction chemotherapy, as well as patients with a relapse of AML oder MDS IB2 after chemotherapy. Patients will receive a combination therapy of ten days of Decitabine and twenty-eigt days of Venetoclax. If hematologic remission is not achieved after one cycle of treatment, patients receive a second cycle. After treatment, a follow-up period of 100 days will ensue. The main aim of the trial is the assessment of hematologic remission after combining Venetoclax with a time-dense immediate application of the hypomethylating agent Decitabine after failure of a chemotherapy approach, thus additionally altering backbone treatment modalities from chemotherapy to epigenetic and anti-BCL2 (B-cell lymphoma 2) treatment. A first assessment of safety and feasibility will take place after the treatment of three patients and a second assessment for safety, feasibility and efficacy/futility after nine patients.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of AML according to WHO criteria regardless of subtype, including de novo and transformed MPN and transformed MDS 2. A. Refractory to induction chemotherapy consisting of Daunorubicin+Cytarabin ("3+7") based chemotherapy, including CPX351, including combinations with GemtuzumabOzogamicin or with the FLT3-inhibitors Midostaurin or Quizartinib. This trial defines refractory disease as one of the following: i. ≥20% bone marrow blasts** at day 15*** first cycle of intensive induction chemotherapy ii. ≥5-20% bone marrow blasts** at day 15*** of first cycle of intensive induction chemotherapy in patients, in whom relative blast count reduction as compared to initial diagnosis is ≤50% iii. c) ≥5% bone marrow blasts** at day 28**** of first cycle of induction chemotherapy, or at any point during a second cycle of induction chemotherapy OR 2. B. Relapse of AML/MDS IB2 after chemotherapy (≥5% medullary blasts in bone marrow assessment**) 3. Must be ≥ 18 years at the time of signing the informed consent. 4. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures. 5. Able to adhere to the study visit schedule and other protocol requirements. 6. Patient is fit for aggressive induction chemotherapy and transplantation by assessment of an experienced hematologist 7. No known history of chronic pulmonary disease and absence of dyspnea. Otherwise, documented diffusion lung capacity for carbon monoxide (DLCO) >40% (adjusted for hemoglobin, if available) and FEV1/FVC >50% 8. Subject (male or female (FCBP))1 is willing to use highly effective birth control methods during treatment and for 3 months (male) and 6 months (female) after the end of treatment (adequate: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition ofvulation, intrauterine device, intrauterine hormone-releasing system bilateral tubal occlusion, vasectomized partner2 sexual abstinence3). Female subjects who use hormonal contraceptives should also use a barrier method.

1. A FCBP is defined as any female who does not meet the criteria of non-childbearing potential. These are as follows:

   * documented hysterectomy, bilateral oophorectomy (ovarectomy), or bilateral tubal ligation
   * post-menopausal (a practical definition accepts menopause ≥ 1 year without menses with an appropriate clinical profile, e.g. age > 45 years in the absence of hormone replacement therapy (HRT). In questionable cases, the subject must have a follicle stimulating hormone (FSH) value > 40 mIU/ml and an estradiol value < 40pg/ml.
2. Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success
3. In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. 9. All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment. 10. All subjects must agree not to share medication.

   * in bone marrow aspiration cytomorphology, or bone marrow pathology, if aspiration morphology not available or not representative *** time frame of tolerance from day 13 to day 20 ****time frame of tolerance from day 21 to day 42

Exclusion Criteria

1. APL (AML with t (15;17))
2. Not consenting to chemotherapy in general
3. Previous Treatment with allogeneic stem cell transplantation
4. ECOG >3
5. Medical History of hypersensitivity to to the active substances of Venetoclax and Decitabin or to any of the excipients listed in the respective SmPCs
6. Relapsed FLT3-ITD- or FLT3-TKD-mutated patients, who previously responded (CR, CRi, CRh or MLFS) to a regimen containing a FLT3-inhibitor.
7. Women during pregnancy and lactation.
8. Significant active cardiac disease within 6 months prior to the start of study treatment, including:

   * New York Heart Association (NYHA) class III or IV congestive heart failure;
   * Myocardial infarction;
   * Unstable angina and/or stroke;
   * Severe cardiac arrhythmias
   * Left ventricular ejection fraction (LVEF) <40% by ultrasound obtained within 28 days prior to the start of study treatment.
9. Severe obstructive or restrictive ventilation disorder
10. Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. (Note: Evaluation of cerebrospinal fluid (CSF) during screening is only required if there is a clinical suspicion of CNS involvement by leukemia during screening)
11. Active infection, including hepatitis B or hepatitis C antibody or Human Immunodeficiency Virus (HIV) infection, that is uncontrolled prior to first dose of study treatment and may interfere with the study objectives or which could expose the patient to undue risk through the participation in the clinical trial; an infection controlled with an approved antibiotic/ antiviral/ antifungal treatment that is not a strong or moderate CYP3A4 inducer is allowed.
12. Immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding and/or disseminated intravascular coagulation
13. Conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs.
14. Patients with a currently active second malignancy. Patients are not considered to have a currently active malignancy if they have completed therapy and are considered by their physician to be at <30% risk of relapse within one year. However, patients with the following history/concurrent conditions are allowed:

    * Basal or squamous cell carcinoma of the skin;
    * Carcinoma in situ of the cervix;
    * Carcinoma in situ of the breast;
    * Incidental histologic finding of prostate cancer.
15. Receipt of live, attenuated vaccine within 30 days prior to the study inclusion (NOTE: patients, if enrolled, should not receive live vaccine during the study and until 6 months after the therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of hematological remissions | measured after the first and second cycle (each cycle is 28 days)
  Hematologic remission (defined as morphologically leukemia-free state (MLFS), complete remission (CR), complete remission with incomplete hematological recovery (CRi) or complete remission with partial hematological recovery (CRh)) as best response in bone marrow aspiration cytomorphology*) after one or two cycles of Decitabine/Venetoclax.
  * or bone marrow pathology, if aspiration morphology not available, not representative or not judged sufficiently reliable by treating physician

SECONDARY OUTCOMES:
Rate of CTCAEs ≥ Grade 3 | observed during the first and second cycle (each cycle is 28 days) and until day 30 after therapy application
  evaluated by the incidence of CTCAEs ≥ Grade 3
Time to hematopoietic recovery in days | after each chemotherapy treatment cycle (28 days), defined as the time from the start of the cycle until recovery
  hematopoietic recovery defined as absolute neutrophil counts ≥0.5 and ≥1.0 x 109/L; platelets ≥50 and ≥100 x 109/L)
Rate of MRD-negativity (measurable residual disease) | measured at each remission assessment (C1D15, C1D28, C2D28, Follow Up)
  MRD including qPCR for established MRD markers and NGS for exploratory MRD markers is evaluated at each remission assessment
Rate of infectious complications CTCAEs ≥ grade 3 | measured during the first and second cycle and the first 30 days after end of treatment (each cycle is 28 days)
  evaluated by the incidence of infections CTCAEs ≥ grade 3
Time to transplant in days | until day 100 after end of treatment
  defined as days from diagnosis of primary induction failure or relapse to infusion of allogeneic hematopoietic stem cells
Progression-free survival | day 100 after end of treatment
  defined as rate of patients alive without hematological progression at day 100 after end of treatment (and time dependent)
Overall survival | day 100 after end of treatment
  defined as rate of patients alive at day 100 after end of treatment (and time dependent)
Early Mortality | day 30 after start of treatment
  Defined as patients no longer alive at day 30 after start of treatment
Quality of Life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30)) | at screening and at the end of cycle one and two (one cycle is 28 days) and at follow up (day 100 after end of treatment)
  evaluated with the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) at screening, and at the end of cycle one and two, as well as at follow up; scale scores ranging from 0 to 100 with higher scores indicating better outcomes
Hospitalisation days | Day 1 of therapy until day 30 after end of treatment
  Hospitalisation days, defined as days in hospital (days in the outpatient clinic are not counted) from day 1 of therapy until day 30 after end of treatment
ECOG prior to start of conditioning for transplant | between end of treatment and follow up
  ECOG prior to start of conditioning for transplant in all patients who proceed to alloHSCT

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lengerke, Prof., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No